CLINICAL TRIAL: NCT01830946
Title: The Effect of Nighttime Macronutrient Choice and Combined Resistance and High-Intensity Interval Training on Body Composition, Cardiovascular Health, Resting Metabolism, Appetite and Strength in Overweight and Obese Adults
Brief Title: Nighttime Macronutrient Choice and Combined Resistance and High-intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC2011.7210
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Protein; Metabolism; Nighttime eating; Exercise Training
MeSH Terms: conditions — Obesity | interventions — Whey Proteins; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey Protein and Exercise Training (Experimental): This arm involves 4 weeks of consuming a whey protein supplement late in the evening before bed along with combined resistance and high-intensity interval training 3 days per week for 4 weeks (two days of resistance training and one day of high-intensity interval training).
  Interventions: Other: Whey Protein; Other: Combined Resistance and High-Intensity Interval training
- Carbohydrate and Exercise Training (Placebo Comparator): This arm involves 4 weeks of consuming a carbohydrate placebo late in the evening before bed along with combined resistance and high-intensity interval training 3 days per week for 4 weeks (two days of resistance training and one day of high-intensity interval training).
  Interventions: Other: Combined Resistance and High-Intensity Interval training
- Casein Protein and Exercise Training (Experimental): This arm involves 4 weeks of consuming a casein protein supplement late in the evening before bed along with combined resistance and high-intensity interval training 3 days per week for 4 weeks (two days of resistance training and one day of high-intensity interval training).
  Interventions: Other: Combined Resistance and High-Intensity Interval training; Other: Casein Protein

INTERVENTIONS:
Other: Whey Protein — Whey protein will be consumed every night of the week as the last food or caloric beverage prior to sleep in the evening at least two hours after dinner but no more than 30 minutes before bed.
  Arms: Whey Protein and Exercise Training
Other: Combined Resistance and High-Intensity Interval training — Completed 3 d/wk for 4 wks (2 d of Resistance Training (RT) and 1 d of High-Intensity Interval Training (HITT)). RT exercises were chest press, seated row,leg press, shoulder press, leg extension, and leg curl (3 total sets: 2 sets of 10 repetitions and a 3rd set to muscular exhaustion with a load equaling 75-85% of 1-Repetition Maximum(RM)). All exercises and sets were separated by 90-120 sec of rest. HIIT training was completed on commerical cardiovascular equipment and requires subjects to rate their perceived exertion on a scale from 1 to 10 (1= resting quietly, 5= a warm-up level, 10= an all-out exertion). Subjects warmed-up for 2 min at level 5 and increased their exertion each min for 3 min until level 9 is perceived and then recover at level 6 for 1 min. This pattern was repeated 4 times, where the 4th cycle subjects increased their last min of exertion to level 10, followed by 1-min recovery at the initial warm-up level 5.
Other: Casein Protein — Casein protein will be consumed every night of the week as the last food or caloric beverage prior to sleep in the evening at least two hours after dinner but no more than 30 minutes before bed.
  Arms: Casein Protein and Exercise Training

SUMMARY:
Obesity is recognized as a major public health concern because of its link to potential fatal complications arising from metabolic and cardiovascular diseases. Despite many pharmacological advances in this field, lifestyle strategies that emphasize proper nutrient intake and physical activity continue to be the primary strategy for individuals to fight obesity. However, controversy exists regarding the type and timing of exercise and specific nutrient intake to maximize fat loss, muscle gain, and beneficial cardio-metabolic adaptations derived from these lifestyle interventions. Furthermore, limited data exists investigating the impact of nutrient timing at times other than immediately before or after exercise and no studies have examined time-of-day nutritional intake in overweight or obese individuals.In addition, many individuals attempting to improve body composition and cardio-metabolic health are concerned with what food choices are appropriate in the late evening to support positive physiological adaptations. However, research-based information examining this topic is scarce.

The investigators hypothesize that consumption of a protein beverage in the late evening before sleep will improve body composition, cardio-metabolic health, and adaptations to exercise more than an isocaloric placebo beverage. The investigators also hypothesize that the different digestion and absorption kinetics of whey and casein proteins will elicit different effects on the measures variables.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of consumption of a protein beverage in the late evening before sleep along with the combination of resistance and high-intensity interval training on improving body composition, muscle strength and overall health compared to a carbohydrate placebo beverage in overweight and obese individuals. Specifically, we will be measuring heart rate, blood pressure, body composition, resting metabolism, maximal strength,cardiovascular function, hormones levels, blood lipid profile, appetite, mood state, and dietary intake. Specific aims of the study are:

To determine if acute ingestion of a liquid ready-to-drink protein supplement (30g whey or casein protein per serving) consumed in the late evening before sleep will alter the physiological milieu to favor anabolism and alter lipolysis and fat oxidation more than the carbohydrate placebo (34g of maltodextrin per serving).

To determine if 4 weeks of daily protein supplementation (same supplement as above) in the late evening along with 3 days of exercise training per week will improve body composition, blood lipid profile, strength, cardiovascular risk profile more than a placebo beverage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Sedentary(exercises <2 days per week for more than 40 minutes per session within the past 6 months)
* overweight or obese (BMI ≥ 25)

Exclusion Criteria:

* Those that exercise for more than 2 days per week for more than 40 minutes per session (within the past 6 months),
* Those that have uncontrolled hypertension (Blood Pressure (BP)>160/100 mmHg)
* Those that take BP medications
* Those diagnosed cardiovascular disease
* Those diagnosed with stroke
* Those diagnosed with diabetes
* Those diagnosed with thyroid dysfunction
* Those diagnosed with kidney dysfunction
* Those with any musculoskeletal complications that would impede exercise
* Those that smoke heavily (>20 cigarettes per day)
* Those that take cholesterol medication
* Those that take nutritional supplements (except for a multivitamin)
* Those with any allergies to milk products

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Body Composition | 4 weeks
  Measuring fat mass and lean mass from dual-energy x-ray absorptiometry.
Metabolism | 4 weeks
  Measured using indirect calorimetry, a non-invasive test that involves lying down on a padded table for 30-minutes with a mouth piece and nose clip

SECONDARY OUTCOMES:
Blood biomarkers | 4 weeks
  Under sterile conditions 20 milliliters of blood was drawn from a forearm antecubital vein and analyzed for blood biomarkers.
Arterial Stiffness | 4 weeks
  Measured using pulse wave velocity of the aorta, systemic, and legs
Appetite | 4 weeks
  Measured by a visual analog scale
Strength | 4 weeks
  Assessed by having the subject progressed towards the maximum weight that they can lift 1-time through a full range of motion and all attempts and will be supervised by trained personnel

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ormsbee, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Ormsbee MJ, Kinsey AW, Eddy WR, Madzima TA, Arciero PJ, Figueroa A, Panton LB. The influence of nighttime feeding of carbohydrate or protein combined with exercise training on appetite and cardiometabolic risk in young obese women. Appl Physiol Nutr Metab. 2015 Jan;40(1):37-45. doi: 10.1139/apnm-2014-0256. PMID 25409324
- [Derived] Figueroa A, Wong A, Kinsey A, Kalfon R, Eddy W, Ormsbee MJ. Effects of milk proteins and combined exercise training on aortic hemodynamics and arterial stiffness in young obese women with high blood pressure. Am J Hypertens. 2014 Mar;27(3):338-44. doi: 10.1093/ajh/hpt224. Epub 2013 Dec 3. PMID 24300595